CLINICAL TRIAL: NCT01066871
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Phase II Trial to Investigate the Efficacy and Safety of Weekly Intra-articular (i.a.) Injections of 10, 30, and 100 µg of AS902330 for Three Consecutive Weeks in Patients With Acute Cartilage Injury of the Knee
Brief Title: Sprifermin (AS902330) in Cartilage Injury Repair (CIR)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was discontinued due to low recruitment.
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMR700692_003
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Results first posted 2016-03-23 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-02

CONDITIONS: Isolated Cartilage Injury of the Knee
Keywords: Knee cartilage injury; fibroblast growth factor 18; FGF18
MeSH Terms: interventions — fibroblast growth factor 18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sprifermin (AS902330) 10 mcg (Experimental)
  Interventions: Drug: Sprifermin (AS902330) 10 mcg
- Sprifermin (AS902330) 30 mcg (Experimental)
  Interventions: Drug: Sprifermin (AS902330) 30 mcg
- Sprifermin (AS902330) 100 mcg (Experimental)
  Interventions: Drug: Sprifermin (AS902330) 100 mcg
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sprifermin (AS902330) 10 mcg — Sprifermin (AS902330) will be administered at a dose of 10 microgram (mcg) as intra-articular injection once every week for 3 consecutive weeks.
  Arms: Sprifermin (AS902330) 10 mcg
Drug: Sprifermin (AS902330) 30 mcg — Sprifermin (AS902330) will be administered at a dose of 30 mcg as intra-articular injection once every week for 3 consecutive weeks.
  Arms: Sprifermin (AS902330) 30 mcg
Drug: Sprifermin (AS902330) 100 mcg — Sprifermin (AS902330) will be administered at a dose of 100 mcg as intra-articular injection once every week for 3 consecutive weeks.
  Arms: Sprifermin (AS902330) 100 mcg
Other: Placebo — Placebo matched to sprifermin (AS902330) will be administered as intra-articular injection once every week for 3 consecutive weeks.
  Arms: Placebo

SUMMARY:
Several people all over the world suffer from cartilage injuries in the knee. Symptoms include pain, joint swelling, and loss of function. Without repair, cartilage injury may ultimately lead to osteoarthritis (OA). Natural healing is poor, and to date treatment is available only for deep cartilage defects involving also the underlying bone. A promising candidate for drug treatment of cartilage injury is sprifermin (AS902330), a recombinant form of the human fibroblast growth factor (FGF) 18.

So far, the drug has been used in subjects with different stages of knee OA in two ongoing studies without emerging safety issues following single and multiple intra-articular injections of ascending doses. However, OA represents late-stage cartilage injury, where repair might be difficult due to diffuse damage, reduced responsiveness of the cartilage, and/or the involvement of other joint structures.

This clinical trial is meant to provide the proof of concept and to identify an efficacious dose of sprifermin (AS902330) for the treatment of adult subjects with acute cartilage injuries of the knee. The first subject for this trial was treated on the 19th of April 2010.

ELIGIBILITY:
Inclusion Criteria:

* Acute cartilage lesion of ICRS grade 2 to 4 at the femoral condyle of the knee (= target knee)
* Age: 18 to 45 years
* Sex: male or female. Women of childbearing potential (that is, all female subjects after puberty unless they are post-menopausal for at least 2 years or surgically sterile) must have negative serum and urine pregnancy tests at screening and Visit 1, respectively, and must use a highly effective method of contraception.
* History of pain and effusion of the target knee post-injury
* Injury within 4 to 12 weeks prior to 1st treatment with investigational medicinal product (IMP)
* Written informed consent prior to any trial-related activity

Exclusion Criteria:

* Personal medical history of osteoarthritis OA in either knee
* Any previous surgery on the target knee
* History of swelling of the target knee along with pain on weight-bearing, or arthroscopy for diagnostic purposes during the 12 months preceding injury
* Corticosteroid (intra-articular) injection into the target knee during the preceding 12 months
* Any other intra-articular injection into the target knee during the preceding 3 months
* Any concurrent injury (for example, arthrolith, anterior cruciate ligament rupture, meniscus tear) of the target knee requiring surgical intervention
* OA or any pre-existing cartilage damage in the target knee, as revealed by MRI
* Legal incapacity or limited legal capacity
* Subjects who are imprisoned or institutionalized by regulatory or court order
* Pregnancy or lactation
* Participation in another clinical trial within the past 30 days
* Any condition or findings in the medical history or in the pre-trial assessments that in the opinion of the Investigator constitutes a risk or contraindication for participation in the trial or that could interfere with the trial objectives, conduct or evaluation
* Known hypersensitivity to the trial treatment or diluents
* Significant renal or hepatic impairment, as indicated by: Aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase (ALP) greater than (>) 3 times the upper limit of normal (ULN); total bilirubin >1.5 times ULN (except in case of Gilbert's syndrome); creatinine >1.5 times ULN; hemoglobin less than (<5.5) millimole per liter (mmol/L), white blood cell count (WBC) <2.5 * 10^9 per liter, or platelets <75 *10^9 per liter)
* Any suspicion of intra-articular infection
* Any known active infections that may compromise the immune system such as human immunodeficiency virus (HIV), Hepatitis B or C infection
* History of sarcoma and/or of other active malignancy within five years, except adequately treated basal cell or squamous cell carcinoma of the skin
* Open growth plate, as revealed by MRI
* Diagnostic arthroscopy after injury and within 4 weeks prior to treatment start

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2010-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Please contact the Merck KGaA Communication Center, Darmstadt, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Sprifermin (AS902330) 10 mcg: Sprifermin (AS902330) was administered at a dose of 10 microgram (mcg) as intra-articular injection once every week for 3 consecutive weeks.
- Sprifermin (AS902330) 30 mcg: Sprifermin (AS902330) was administered at a dose of 30 mcg as intra-articular injection once every week for 3 consecutive weeks.
- Sprifermin (AS902330) 100 mcg: Sprifermin (AS902330) was administered at a dose of 100 mcg as intra-articular injection once every week for 3 consecutive weeks.
- Placebo: Placebo matched to sprifermin (AS902330) was administered as intra-articular injection once every week for 3 consecutive weeks.
Period: Overall Study
Arm/Group | Sprifermin (AS902330) 10 mcg | Sprifermin (AS902330) 30 mcg | Sprifermin (AS902330) 100 mcg | Placebo
Started | 20 | 18 | 18 | 18
Completed | 16 | 13 | 12 | 13
Not Completed | 4 | 5 | 6 | 5
Not completed — Lost to Follow-up | 0 | 2 | 2 | 0
Not completed — Protocol Violation | 1 | 0 | 3 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 0
Not completed — Other | 0 | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Population: The intention-to-treat (ITT) population included all participants randomized to a trial treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sprifermin (AS902330) 10 mcg | Sprifermin (AS902330) 30 mcg | Sprifermin (AS902330) 100 mcg | Placebo | Total
Number analyzed (Participants) | 20 | 18 | 18 | 18 | 74
Age, Customized [Number; unit: participants]
  Less than (<) 40 years | 16 | 15 | 14 | 16 | 61
  Greater than or equal to (>=) 40 years | 4 | 3 | 4 | 2 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 7 | 3 | 20
  Male | 15 | 13 | 11 | 15 | 54

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Cartilage Defect Volume at Month 12
Description: Percent change in cartilage defect volume was calculated based on central magnetic resonance imaging (MRI): (volume at Month 12 minus volume at baseline)*100/volume at baseline.
Time Frame: Baseline, Month 12
Population: The modified intent-to-treat (mITT) analysis set included all participants from the ITT analysis set who had at least 1 post-treatment magnetic resonance imaging assessment. "N" (number of participants analyzed) signifies the participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Sprifermin (AS902330) 10 mcg: Sprifermin (AS902330) was be administered at a dose of 10 microgram (mcg) as intra-articular injection once every week for 3 consecutive weeks.
Arm/Group | Sprifermin (AS902330) 10 mcg | Sprifermin (AS902330) 30 mcg | Sprifermin (AS902330) 100 mcg | Placebo
Number analyzed (Participants) | 16 | 14 | 15 | 16
Percent change | -14.4 (27.17) | -17.8 (29.24) | -12.0 (34.80) | -17.0 (26.65)

2. Secondary Outcome: Percent Change From Baseline in Cartilage Defect Volume and Cartilage Defect Thickness in the Target Knee at Months 3 and 6
Description: Percent change in cartilage defect volume and cartilage defect thickness at Months 3 and 6 based on central MRI was calculated as: ([volume or thickness at Months 3 and 6 minus volume or thickness at baseline, respectively]*100)/volume or thickness at baseline.
Time Frame: Baseline, Months 3 and 6
Population: The mITT analysis set included all participants from the ITT analysis set who had at least 1 post-treatment magnetic resonance imaging assessment. "n" signifies the participants who were evaluable for this outcome measure for each group, respectively.
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- AS902330 10 mcg: AS902330 was administered at a dose of 10 microgram (mcg) as intra-articular injection once every week for 3 consecutive weeks.
- AS902330 30 mcg: AS902330 was administered at a dose of 30 mcg as intra-articular injection once every week for 3 consecutive weeks.
- AS902330 100 mcg: AS902330 was administered at a dose of 100 mcg as intra-articular injection once every week for 3 consecutive weeks.
- Placebo: Placebo matched to sprifermin AS902330 was administered as intra-articular injection once every week for 3 consecutive weeks.
Arm/Group | AS902330 10 mcg | AS902330 30 mcg | AS902330 100 mcg | Placebo
Number analyzed (Participants) | 19 | 16 | 17 | 17
Percent change
  Volume: Month 3 (n=18, 16, 17, 17) | 3.097 (24.7727) | -1.596 (22.6831) | -2.054 (28.3639) | -3.307 (12.3879)
  Volume: Month 6 (n=17, 15, 17, 16) | 0.922 (28.8298) | -11.118 (32.3251) | -7.518 (32.6967) | -6.792 (27.8652)
  Thickness: Month 3 (n=18, 16, 17, 17) | 3.126 (9.7969) | -1.969 (9.2075) | -1.327 (16.4475) | -0.810 (10.9976)
  Thickness: Month 6 (n=17, 15, 17, 16) | 3.461 (11.7686) | -3.184 (14.1109) | -5.439 (16.1866) | -3.106 (14.1901)

3. Secondary Outcome: Change From Baseline in Cartilage Defect Volume in the Target Knee at Months 3, 6 and 12
Description: The change in cartilage defect volume at Months 3, 6 and 12 based on central MRI was calculated as volume at Months 3, 6 and 12 minus volume at baseline, respectively.
Time Frame: Baseline, Months 3, 6 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: microliter
Arm/Group | Sprifermin (AS902330) 10 mcg | Sprifermin (AS902330) 30 mcg | Sprifermin (AS902330) 100 mcg | Placebo
Number analyzed (Participants) | 19 | 16 | 17 | 17
microliter
  Baseline (n=19, 16, 17, 17) | 130.689 (83.7032) | 190.354 (130.5796) | 158.125 (131.2277) | 128.982 (116.9241)
  Change at Month 3 (n=18, 16, 17, 17) | 1.682 (30.2235) | -5.588 (21.5146) | -9.630 (40.2382) | -7.439 (13.7056)
  Change at Month 6 (n=17, 15, 17, 16) | -0.540 (34.6432) | -29.830 (47.7638) | -23.469 (59.1138) | -14.511 (28.3908)
  Change at Month 12 (n=16, 14, 15, 16) | -13.492 (40.8876) | -35.800 (37.0570) | -39.658 (80.5121) | -25.188 (36.1098)

4. Secondary Outcome: Change From Baseline in Cartilage Defect Thickness in the Target Knee at Months 3, 6 and 12
Description: The change in cartilage defect thickness at Months 3, 6 and 12 based on central MRI was calculated as thickness at Months 3, 6 and 12 minus thickness at baseline, respectively.
Time Frame: Baseline, Months 3, 6 and 12
Population: The modified intent-to-treat (mITT) analysis set included all participants from the ITT analysis set who had at least 1 post-treatment magnetic resonance imaging assessment. "n" signifies the participants who were evaluable for this outcome measure for each group, respectively.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Sprifermin (AS902330) 10 mcg | Sprifermin (AS902330) 30 mcg | Sprifermin (AS902330) 100 mcg | Placebo
Number analyzed (Participants) | 19 | 16 | 17 | 17
millimeter
  Baseline (n=19, 16, 17, 17) | 1.598 (0.5550) | 1.903 (0.5685) | 1.758 (0.4901) | 1.641 (0.5625)
  Change at Month 3 (n=18, 16, 17, 17) | 0.028 (0.1441) | -0.029 (0.1847) | -0.046 (0.2544) | -0.005 (0.1633)
  Change at Month 6 (n=17, 15, 17, 16) | 0.041 (0.1873) | -0.066 (0.2887) | -0.131 (0.2441) | -0.043 (0.2088)
  Change at Month 12 (n=16, 14, 15, 16) | -0.058 (0.2648) | -0.101 (0.2318) | -0.176 (0.3274) | -0.179 (0.1661)

5. Secondary Outcome: Number of Participants With Response to Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) Sub-scales
Description: MOCART scoring system (comprising 9 variables) was used to describe the morphology & signal intensity of the repair tissue following MRI -degree of defect repair [DDR] score 0 (subchondral bone exposed) to 20 (complete repair); integration to the border zone [IBZ] score 0 (> 50% of length of repair tissue) to 15 (complete integration to border zone);surface of repair tissue [SRT] score 0 (>50% surface repair tissue/total degradation) to 10(surface intact);structure of repair tissue [StRT] score 0(inhomogenous/cleft formation) to 5 (homogenous);signal intensity [T2] Mapping Sequence [T2MS] and Hi-Res Sagittal Pharmacodynamic Sequence [Hi-Res SPS] score 0 (marked hyper intense for T2MS and hypo intense for Hi-Res SPS) to 15 (iso intense); subchondral lamina,subchondral bone score 0 (not impact) to 5 (intact);adhesions & effusion score 0 (yes) and 5 (no). Higher values represent more favorable outcome of repair.
Time Frame: Months 3 (M3), 6 (M6) and 12 (M12)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Sprifermin (AS902330) 10 mcg | Sprifermin (AS902330) 30 mcg | Sprifermin (AS902330) 100 mcg | Placebo
Number analyzed (Participants) | 19 | 16 | 17 | 17
participants
  M3, DDR, Complete (n=4, 4, 3, 6) | 0 | 1 | 0 | 0
  M3, DDR, Hypertrophy (n=4, 4, 3, 6) | 0 | 0 | 0 | 0
  M3, DDR, incomplete >50% (n=4, 4, 3, 6) | 1 | 1 | 2 | 1
  M3, DDR, incomplete<50% (n=4, 4, 3, 6) | 3 | 2 | 1 | 5
  M3, DDR, subchondral bone exposed (n=4, 4, 3, 6) | 0 | 0 | 0 | 0
  M6, DDR, Complete (n=3, 5, 3, 6) | 0 | 1 | 0 | 0
  M6, DDR, Hypertrophy (n=3, 5, 3, 6) | 0 | 0 | 0 | 0
  M6, DDR, incomplete >50% (n=3, 5, 3, 6) | 1 | 1 | 2 | 0
  M6, DDR, incomplete<50% (n=3, 5, 3, 6) | 2 | 3 | 1 | 6
  M6, DDR, subchondral bone exposed (n=3, 5, 3, 6) | 0 | 0 | 0 | 0
  M12, DDR, Complete (n=4, 8, 2, 5) | 0 | 1 | 0 | 0
  M12, DDR, Hypertrophy (n=4, 8, 2, 5) | 0 | 0 | 0 | 0
  M12, DDR, incomplete >50% (n=4, 8, 2, 5) | 3 | 1 | 1 | 0
  M12, DDR, incomplete<50% (n=4, 8, 2, 5) | 1 | 6 | 1 | 5
  M12, DDR, subchondral bone exposed (n=4, 8, 2, 5) | 0 | 0 | 0 | 0
  M3, IBZ, Complete (n=1, 1, 0, 2) | 1 | 1 | 0 | 2
  M3, IBZ, Incomplete (split-like) (n=1, 1, 0, 2) | 0 | 0 | 0 | 0
  M3,IBZ,Defect visible<50% repair tissue(n=1,1,0,2) | 0 | 0 | 0 | 0
  M3,IBZ,Defect visible>50% repair tissue(n=1,1,0,2) | 0 | 0 | 0 | 0
  M6, IBZ, Complete (n=1, 2, 0, 2) | 1 | 2 | 0 | 2
  M6, IBZ, Incomplete (split-like) (n=1, 2, 0, 2) | 0 | 0 | 0 | 0
  M6,IBZ,Defect visible<50% repair tissue(n=1,2,0,2) | 0 | 0 | 0 | 0
  M6,IBZ,Defect visible>50% repair tissue(n=1,2,0,2) | 0 | 0 | 0 | 0
  M12, IBZ, Complete (n=1, 2, 0, 1) | 1 | 2 | 0 | 1
  M12, IBZ, Incomplete (split-like) (n=1, 2, 0, 1) | 0 | 0 | 0 | 0
  M12,IBZ,Defect visible<50% repair tissue(n=1,2,0,1 | 0 | 0 | 0 | 0
  M12,IBZ,Defect visible>50% repair tissue(n=1,2,0,1 | 0 | 0 | 0 | 0
  M3, SRT, surface intact (n=1, 1, 0, 2) | 1 | 1 | 0 | 2
  M3, SRT, surface damaged < 50% (n=1, 1, 0, 2) | 0 | 0 | 0 | 0
  M3, SRT, surface damaged > 50% (n=1, 1, 0, 2) | 0 | 0 | 0 | 0
  M6, SRT, surface intact (n=1, 2, 0, 2) | 1 | 2 | 0 | 2
  M6, SRT, surface damaged <50% (n=1, 2, 0, 2) | 0 | 0 | 0 | 0
  M6, SRT, surface damaged > 50% (n=1, 2, 0, 2) | 0 | 0 | 0 | 0
  M12, SRT, surface intact (n=1, 2, 0, 1) | 1 | 2 | 0 | 1
  M12, SRT, surface damaged <50% (n=1, 2, 0, 1) | 0 | 0 | 0 | 0
  M12, SRT, surface damaged > 50% (n=1, 2, 0, 1) | 0 | 0 | 0 | 0
  M3, StRT, Homogeneous (n=4, 3, 0, 4) | 4 | 3 | 0 | 4
  M3, StRT, Inhomogenous (n=4, 3, 0, 4) | 0 | 0 | 0 | 0
  M6, StRT, Homogeneous (n=3, 4, 0, 3) | 3 | 3 | 0 | 3
  M6, StRT, Inhomogenous (n=3, 4, 0, 3) | 0 | 1 | 0 | 0
  M12, StRT, Homogeneous (n=3, 4, 0, 2) | 3 | 3 | 0 | 2
  M12, StRT, Inhomogenous(n=3, 4, 0, 2) | 0 | 1 | 0 | 0
  M3, T2MS, Isointense (n=5, 4, 3, 6) | 5 | 4 | 3 | 6
  M3, T2MS, Moderately hyperintense (n=5, 4, 3, 6) | 0 | 0 | 0 | 0
  M3, T2MS, Markedly hyperintense (n=5, 4, 3, 6) | 0 | 0 | 0 | 0
  M6, T2MS, Isointense (n=4, 5, 3, 6) | 4 | 5 | 3 | 6
  M6, T2MS, Moderately hyperintense (n=4, 5, 3, 6) | 0 | 0 | 0 | 0
  M6, T2MS, Markedly hyperintense (n=4, 5, 3, 6) | 0 | 0 | 0 | 0
  M12, T2MS, Isointense (n=4, 8, 2, 5) | 4 | 8 | 2 | 5
  M12, T2MS, Moderately hyperintense (n=4, 8, 2, 5) | 0 | 0 | 0 | 0
  M12, T2MS, Markedly hyperintense (n=4, 8, 2, 5) | 0 | 0 | 0 | 0
  M3, Hi-Res SPS, Isointense (n=5, 4, 3, 6) | 5 | 4 | 3 | 6
  M3, Hi-Res, Moderately hypointense (n=5, 4, 3, 6) | 0 | 0 | 0 | 0
  M3, Hi-Res, Markedly hypointense (n=5, 4, 3, 6) | 0 | 0 | 0 | 0
  M6, Hi-Res SPS, Isointense (n=4, 5, 3, 6) | 4 | 4 | 3 | 6
  M6, Hi-Res, Moderately hypointense (n=4, 5, 3, 6) | 0 | 1 | 0 | 0
  M6, Hi-Res, Markedly hypointense (n=4, 5, 3, 6) | 0 | 0 | 0 | 0
  M12, Hi-Res SPS, Isointense (n=4, 8, 2, 5) | 4 | 6 | 1 | 5
  M12, Hi-Res, Moderately hypointense (n=4, 8, 2, 5) | 0 | 2 | 1 | 0
  M12, Hi-Res, Markedly hypointense (n=4, 8, 2, 5) | 0 | 0 | 0 | 0
  M3, Subchondral Lamina Intact (n=17, 16, 17, 17) | 17 | 16 | 17 | 17
  M3, Subchondral Lamina Not Intact (n=17,16,17,17) | 0 | 0 | 0 | 0
  M6, Subchondral Lamina Intact (n=16, 15, 17, 16) | 16 | 15 | 17 | 16
  M6, Subchondral Lamina Not Intact (n=16,15,17,16) | 0 | 0 | 0 | 0
  M12, Subchondral Lamina Intact (n=15, 14, 15, 16) | 15 | 14 | 15 | 16
  M12,Subchondral Lamina Not Intact (n=15,14,15,16) | 0 | 0 | 0 | 0
  M3, Subchondral bone Intact (n=18, 16, 17, 17) | 16 | 16 | 17 | 17
  M3, Subchondral bone Not Intact (n=18, 16, 17, 17) | 2 | 0 | 0 | 0
  M6, Subchondral bone Intact (n=17, 15, 17, 16) | 14 | 15 | 16 | 15
  M6, Subchondral bone Not Intact (n=17, 15, 17, 16) | 3 | 0 | 1 | 1
  M12, Subchondral bone Intact (n=16, 14, 15, 16) | 12 | 13 | 14 | 16
  M12, Subchondral bone Not Intact (n=16, 14, 15, 16 | 4 | 1 | 1 | 0
  M3, Adhesions-No (n=2, 3, 1, 2) | 2 | 3 | 1 | 2
  M3, Adhesions-Yes (n=2, 3, 1, 2) | 0 | 0 | 0 | 0
  M6, Adhesions-No (n=3, 3, 1, 3) | 3 | 3 | 1 | 3
  M6, Adhesions-Yes (n=3, 3, 1, 3) | 0 | 0 | 0 | 0
  M12, Adhesions-No (n=2, 5, 1, 2) | 2 | 5 | 1 | 2
  M12, Adhesions-Yes (n=2, 5, 1, 2) | 0 | 0 | 0 | 0
  M3, Effusion-No (n=18, 16, 17, 17) | 5 | 2 | 1 | 3
  M3, Effusion-Yes (n=18, 16, 17, 17) | 13 | 14 | 16 | 14
  M6, Effusion-No (n=17, 15, 17, 16) | 4 | 2 | 3 | 4
  M6, Effusion-Yes (n=17, 15, 17, 16) | 13 | 13 | 14 | 12
  M12, Effusion-No (n=16, 14, 15, 16) | 3 | 4 | 1 | 3
  M12, Effusion-Yes (n=16, 14, 15, 16) | 13 | 10 | 14 | 13

6. Secondary Outcome: Change From Baseline in Boston Leeds Osteoarthritis Knee Score (BLOKS) Sub-scale (Bone Marrow Lesion [BML] Size, Osteophyte Size, Meniscal Extrusion Score [MES], and Meniscal Tear Score [MTS]) Scores at Month 12
Description: The BLOKS scoring system assesses intra-articular regions within the knee according to the following features: BML size, cartilage 1, osteophyte size, synovitis, effusion, meniscal extrusion, and meniscal tear. Change from baseline in summary scores for BML size, osteophyte size, MES, and MTS were reported. Summary scores for BML size range from 0 to 27, for osteophyte size range from 0 to 36, for MES range from 0 to 12, and for MTS range from 0 to 32, with lower scores corresponding to favorable outcomes.
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sprifermin (AS902330) 10 mcg | Sprifermin (AS902330) 30 mcg | Sprifermin (AS902330) 100 mcg | Placebo
Number analyzed (Participants) | 19 | 16 | 17 | 17
units on a scale
  BML: Baseline (n=19, 16, 17, 17) | 1.68 (2.262) | 1.75 (2.933) | 1.24 (1.348) | 1.94 (2.512)
  BML: Change at Month 12(n=16, 14, 15, 16) | -0.69 (2.089) | -1.07 (3.149) | -0.27 (1.033) | -0.88 (1.455)
  Osteophyte: Baseline (n=19, 16, 17, 17) | 0.37 (0.831) | 0.00 (0.000) | 0.88 (1.799) | 0.24 (0.664)
  Osteophyte: Change at Month12 (n=16, 14, 15, 16) | -0.06 (0.250) | 0.07 (0.267) | 0.47 (0.990) | 0.06 (0.250)
  MES: Baseline (n=19, 16, 17, 17) | 0.26 (0.452) | 0.25 (0.577) | 0.47 (0.800) | 0.24 (0.562)
  MES: Change at Month 12 (n=16, 14, 15, 16) | 0.13 (0.342) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  MTS: Baseline (n=19, 16, 17, 17) | 1.05 (1.508) | 0.38 (0.719) | 0.88 (1.219) | 0.53 (0.800)
  MTS: Change at Month 12 (n=16, 14, 15, 16) | 0.13 (0.500) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.365)

7. Secondary Outcome: Number of Participants With Shift From Baseline in BLOKS Sub-Scales (Cartilage 1, Synovitis, Effusion) Scores at Month 12
Description: The BLOKS scoring system assesses intra-articular regions within the knee according to the following features: BML size, cartilage 1, osteophyte size, synovitis, effusion, meniscal extrusion, and meniscal tear. Total number of participants with shift from baseline in various BLOKS sub-scales (cartilage 1 [patella medial, patella lateral, femur medial trochlea, femur lateral trochlea, medial weight bearing femur, lateral weight bearing femur, tibia medial, tibia lateral], synovitis, and effusion) scores at Month 12 were reported.
Time Frame: Month 12
Population: The mITT analysis set included all participants from the ITT analysis set who had at least 1 post-treatment magnetic resonance imaging assessment.
Measure: Number; unit: participants
Arm/Group | Sprifermin (AS902330) 10 mcg | Sprifermin (AS902330) 30 mcg | Sprifermin (AS902330) 100 mcg | Placebo
Number analyzed (Participants) | 19 | 16 | 17 | 17
participants
  Cartilage 1 patella medial | 3 | 1 | 0 | 3
  Cartilage 1 patella lateral | 3 | 1 | 3 | 3
  Cartilage 1 femur medial trochlea | 2 | 1 | 1 | 1
  Cartilage 1 femur lateral trochlea | 3 | 0 | 1 | 1
  Cartilage 1 medial weight bearing femur | 9 | 4 | 2 | 3
  Cartilage 1 lateral weight bearing femur | 2 | 3 | 2 | 2
  Cartilage 1 tibia medial | 0 | 0 | 1 | 1
  Cartilage 1 tibia lateral | 0 | 2 | 2 | 0
  Synovitis | 0 | 1 | 0 | 0
  Effusion | 13 | 11 | 13 | 8

8. Secondary Outcome: Number of Participants With Change From Baseline in International Cartilage Repair Society (ICRS) Grade at Months 6 and 12
Description: The ICRS grading is used to score the amount of cartilage repair and damage. The grades range from 1 to 4 where higher grades indicate more severity of injury. Number of participants with change value of -3, -2, -1, 0, 1, and 2 from baseline in ICRS grade at Months 6 and 12 were reported. Lower change value indicates less severity of injury.
Time Frame: Baseline, Months 6 and 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Sprifermin (AS902330) 10 mcg | Sprifermin (AS902330) 30 mcg | Sprifermin (AS902330) 100 mcg | Placebo
Number analyzed (Participants) | 19 | 16 | 17 | 17
participants
  Month 6: Change value of -3 (n=17, 15, 17, 16) | 0 | 0 | 0 | 0
  Month 6: Change value of -2 (n=17, 15, 17, 16) | 0 | 3 | 1 | 0
  Month 6: Change value of -1 (n=17, 15, 17, 16) | 1 | 6 | 3 | 5
  Month 6: Change value of 0 (n=17, 15, 17, 16) | 13 | 5 | 11 | 10
  Month 6: Change value of 1 (n=17, 15, 17, 16) | 3 | 0 | 1 | 1
  Month 6: Change value of 2 (n=17, 15, 17, 16) | 0 | 1 | 1 | 0
  Month 12: Change value of -3 (n=16, 14, 15, 16) | 0 | 1 | 0 | 0
  Month 12: Change value of -2 (n=16, 14, 15, 16) | 0 | 1 | 1 | 0
  Month 12: Change value of -1 (n=16, 14, 15, 16) | 2 | 5 | 3 | 4
  Month 12: Change value of 0 (n=16, 14, 15, 16) | 12 | 6 | 9 | 11
  Month 12: Change value of 1 (n=16, 14, 15, 16) | 2 | 0 | 2 | 1
  Month 12: Change value of 2 (n=16, 14, 15, 16) | 0 | 1 | 0 | 0

9. Secondary Outcome: Change From Baseline in Knee Injury and Osteoarthritis Outcome Score (KOOS) Sub-scale Scores and International Knee Documentation Committee (IKDC) Score at Months 3, 6 and 12
Description: The KOOS is a knee-specific self-administered questionnaire that assesses symptoms and problems associated with knee injury and osteoarthritis. It consists of 42 items grouped into 5 sub-scales: symptoms, pain, function in daily living (FDL), function in sports and recreation activities (FSRA), and quality of life (QoL). Sub-scale scores range from 0-100, with 0 representing extreme knee problems and 100 no knee problems. The IKDC consists of 19 items to summarize symptoms such as highest level of activity without significant pain, frequency and severity of pain scales, stiffness and swelling, highest levels of activity without significant swelling or giving way, knee lock or catch, highest level of activity that can be performed on a regular basis, effect of knee on ability to perform set tasks, knee function prior to injury, and current knee function. The IKDC scores range from 0-100 where high score represents high levels of function.
Time Frame: Baseline, Months 3, 6 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sprifermin (AS902330) 10 mcg | Sprifermin (AS902330) 30 mcg | Sprifermin (AS902330) 100 mcg | Placebo
Number analyzed (Participants) | 19 | 16 | 17 | 17
units on a scale
  KOOS Symptoms: Baseline (n=19, 16, 17, 17) | 68.80 (16.955) | 67.63 (20.432) | 59.66 (17.024) | 67.65 (21.297)
  KOOS Symptoms:Change at Month 3(n=19, 16, 17, 17) | 14.10 (16.940) | 12.95 (20.982) | 21.01 (13.236) | 17.02 (23.095)
  KOOS Symptoms: Change at Month 6(n=18, 16, 17, 17) | 17.26 (18.385) | 17.19 (16.864) | 26.47 (11.012) | 22.27 (23.975)
  KOOS Symptoms: Change at Month 12(n=17, 14, 16,16) | 12.61 (20.208) | 17.86 (17.994) | 29.91 (14.219) | 26.12 (23.464)
  KOOS Pain: Baseline (n=19, 16, 17, 17) | 65.20 (19.074) | 67.01 (23.282) | 56.70 (20.672) | 65.20 (22.569)
  KOOS Pain: Change at Month 3 (n=19, 16, 17, 17) | 16.23 (19.162) | 18.75 (18.799) | 24.02 (20.197) | 24.02 (25.852)
  KOOS Pain: Change at Month 6 (n=18,16,17,17) | 19.44 (21.810) | 22.40 (19.496) | 26.63 (16.169) | 27.29 (25.839)
  KOOS Pain: Change at Month 12 (n=17, 14, 16, 16) | 16.99 (21.603) | 18.06 (19.543) | 31.60 (14.868) | 28.47 (24.163)
  KOOS FDL: Baseline (n=19, 16, 17, 17) | 69.89 (18.053) | 74.17 (19.969) | 64.01 (20.694) | 73.83 (24.326)
  KOOS FDL: Change at Month 3 (n=19, 16, 17, 17) | 16.95 (18.630) | 14.25 (15.809) | 21.80 (19.302) | 20.80 (25.123)
  KOOS FDL: Change at Month 6 (n=18, 16, 17, 17) | 18.14 (18.690) | 17.56 (16.883) | 25.09 (15.637) | 23.05 (25.792)
  KOOS FDL: Change at Month 12 (n=17, 14, 16, 16) | 16.70 (20.370) | 14.92 (19.199) | 28.22 (16.183) | 24.75 (25.689)
  KOOS FSRA: Baseline (n=18, 16, 17, 16) | 38.06 (24.920) | 46.25 (23.488) | 38.82 (18.416) | 39.38 (25.747)
  KOOS FSRA: Change at Month 3 (n=18, 16, 17, 16) | 22.78 (27.074) | 25.94 (22.746) | 27.06 (25.924) | 38.44 (28.619)
  KOOS FSRA: Change at Month 6 (n=17, 16, 17, 16) | 27.94 (26.224) | 32.19 (23.307) | 31.47 (23.767) | 42.81 (29.550)
  KOOS FSRA: Change at Month 12 (n=16, 14, 16, 15) | 24.38 (28.336) | 32.05 (30.070) | 40.94 (21.926) | 50.33 (29.669)
  KOOS QoL: Baseline (n=19, 16, 17, 17) | 41.45 (25.277) | 41.41 (14.591) | 34.19 (15.643) | 40.07 (19.398)
  KOOS QoL: Change at Month 3 (n=19, 16, 17, 17) | 9.54 (24.149) | 17.19 (18.042) | 16.54 (23.064) | 23.16 (25.842)
  KOOS QoL: Change at Month 6 (n=18, 16, 17, 17) | 13.89 (26.129) | 23.44 (20.091) | 23.53 (17.888) | 27.94 (28.821)
  KOOS QoL: Change at Month 12 (n=17, 14, 16, 16) | 12.13 (27.729) | 16.52 (23.206) | 29.69 (17.002) | 41.41 (28.401)
  IKDC Score: Baseline (n=19, 16, 17, 17) | 52.753 (18.8009) | 50.431 (12.1996) | 46.045 (15.2838) | 55.646 (19.0396)
  IKDC Score: Change at Month 3 (n=19, 16, 16, 17) | 16.999 (16.6813) | 23.563 (13.5872) | 25.790 (19.6412) | 25.152 (20.1268)
  IKDC Score: Change at Month 6 (n=18, 16, 17, 16) | 21.711 (19.4701) | 28.664 (15.2400) | 30.494 (18.9965) | 27.658 (22.8095)
  IKDC Score: Change at Month 12 (n=17, 14, 16, 16) | 20.284 (21.2408) | 25.944 (17.6274) | 31.787 (19.1616) | 32.184 (23.3421)

10. Secondary Outcome: Number of Participants With Global Evaluation of Treatment Benefit
Description: Participants were asked to evaluate and rate the treatment benefit as poor, fair, good, very good or excellent.
Time Frame: Months 3, 6 and 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Sprifermin (AS902330) 10 mcg | Sprifermin (AS902330) 30 mcg | Sprifermin (AS902330) 100 mcg | Placebo
Number analyzed (Participants) | 19 | 16 | 17 | 17
participants
  Poor: Month 3 (n= 19, 16, 17, 17) | 1 | 1 | 0 | 1
  Fair: Month 3 (n= 19, 16, 17, 17) | 3 | 1 | 0 | 3
  Good: Month 3 (n= 19, 16, 17, 17) | 9 | 6 | 3 | 4
  Very Good: Month 3 (n= 19, 16, 17, 17) | 4 | 5 | 10 | 2
  Excellent: Month 3 (n= 19, 16, 17, 17) | 2 | 3 | 4 | 7
  Poor: Month 6 (n= 18, 16, 17, 17) | 0 | 0 | 0 | 1
  Fair: Month 6 (n= 18, 16, 17, 17) | 3 | 0 | 0 | 2
  Good: Month 6 (n= 18, 16, 17, 17) | 7 | 9 | 5 | 6
  Very Good: Month 6 (n= 18, 16, 17, 17) | 5 | 4 | 9 | 2
  Excellent: Month 6 (n= 18, 16, 17, 17) | 3 | 3 | 3 | 6
  Poor: Month 12 (n= 17, 14, 16, 16) | 0 | 0 | 0 | 0
  Fair: Month 12 (n= 17, 14, 16, 16) | 2 | 0 | 0 | 0
  Good: Month 12 (n= 17, 14, 16, 16) | 6 | 3 | 3 | 6
  Very Good: Month 12 (n= 17, 14, 16, 16) | 7 | 5 | 7 | 6
  Excellent: Month 12 (n= 17, 14, 16, 16) | 2 | 6 | 6 | 4

11. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Local TEAEs, Systemic TEAEs, TEAEs Leading to Discontinuation and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An SAE is an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAEs are those AEs that either started or worsened in severity on or after the date of first dose of study drug and on or before Month 12. Local TEAEs are those only related to the target knee. Systemic TEAEs are those that are related to other parts of the body.
Time Frame: Baseline up to Month 12
Population: Safety analysis set included all participants who received at least 1 dose of trial treatment and who had at least 1 post injection safety assessment.
Measure: Number; unit: participants
Arm/Group | Sprifermin (AS902330) 10 mcg | Sprifermin (AS902330) 30 mcg | Sprifermin (AS902330) 100 mcg | Placebo
Number analyzed (Participants) | 19 | 18 | 18 | 19
participants
  TEAEs | 10 | 11 | 12 | 14
  Local TEAEs | 9 | 8 | 11 | 11
  Systemic TEAEs | 6 | 7 | 5 | 7
  TEAEs Leading to Discontinuation | 0 | 0 | 0 | 1
  SAEs | 1 | 0 | 2 | 0

12. Secondary Outcome: Number of Participants With Acute Inflammatory Reactions
Description: Acute inflammatory reaction (AIR) is defined as an increase of pain by 30 millimeter (mm) on a 100 mm visual analog scale (VAS) associated with a subject-reported synovial fluid effusion within 3 days following intra-articular injection.
Time Frame: Baseline up to Month 12
Population: Safety analysis set included all participants who received at least 1 dose of trial treatment and who had at least 1 post injection safety assessment. "N" (number of participants analyzed) signifies the participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Sprifermin (AS902330) 10 mcg | Sprifermin (AS902330) 30 mcg | Sprifermin (AS902330) 100 mcg | Placebo
Number analyzed (Participants) | 14 | 14 | 15 | 12
participants | 4 | 0 | 7 | 2

13. Secondary Outcome: Number of Participants With Binding Antibodies (BAbs) and Neutralizing Antibodies (NAbs) to Fibroblast Growth Factor 18 (FGF18)
Description: Number of participants with BAbs and NAbs to FGF18 at Week 1 (pre-dose), Week 2 (pre-dose), Week 4, Months 3 and 12 were reported.
Time Frame: Week 1 (pre-dose), Week 2 (pre-dose), Week 4, Months 3 and 12
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Sprifermin (AS902330) 10 mcg | Sprifermin (AS902330) 30 mcg | Sprifermin (AS902330) 100 mcg | Placebo
Number analyzed (Participants) | 19 | 18 | 18 | 19
participants
  BAbs: Pre-dose Week 1 | 1 | 2 | 1 | 1
  BAbs: Pre-dose Week 2 | 1 | 3 | 1 | 1
  BAbs: Week 4 | 1 | 3 | 1 | 1
  BAbs: Month 3 | 1 | 3 | 0 | 1
  BAbs: Month 12 | 1 | 1 | 0 | 1
  NAbs: Pre-dose Week 1 | 1 | 1 | 1 | 1
  NAbs: Pre-dose Week 2 | 1 | 2 | 1 | 1
  NAbs: Week 4 | 1 | 2 | 1 | 1
  NAbs: Month 3 | 1 | 2 | 0 | 1
  NAbs: Month 12 | 1 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Baseline Up to Month 12
Description: Safety analysis set included all participants who received at least 1 dose of trial treatment and who had at least 1 post injection safety assessment. One participant randomized to sprifermin (AS902330) 10 mcg group actually received placebo treatment, and therefore was included in placebo group for safety analysis.
Arm/Group | Sprifermin (AS902330) 10 mcg | Sprifermin (AS902330) 30 mcg | Sprifermin (AS902330) 100 mcg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/18 | 2/18 | 0/19
Other Adverse Events (participants affected / at risk) | 10/19 | 11/18 | 13/18 | 15/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sprifermin (AS902330) 10 mcg (N=19) | Sprifermin (AS902330) 30 mcg (N=18) | Sprifermin (AS902330) 100 mcg (N=18) | Placebo (N=19)
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sprifermin (AS902330) 10 mcg (N=19) | Sprifermin (AS902330) 30 mcg (N=18) | Sprifermin (AS902330) 100 mcg (N=18) | Placebo (N=19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 5 | 3
Joint crepitation (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 6 | 4 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 2 | 0 | 2
Influenza (Infections and infestations) | 0 | 1 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 3 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 2 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gingival inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 0 | 1
Blood creatine increased (Investigations) | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 3 | 0
Injection site joint pain (General disorders) | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Tachycardia paroxysmal (Cardiac disorders) | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Eye inflammation (Eye disorders) | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was discontinued due to low recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor can with reasonable grounds require changes to the communication which do not change the scientific statement or neutrality of the communication.